CLINICAL TRIAL: NCT02624167
Title: A Phase IIA, Prospective, Randomized, Double-blind, Multiple-dose Study of NW-3509A in Chronic Schizoprhenia Patients Not Responding to Their Current Anti-psychotic Medication
Brief Title: A Study to Determine the Safety, Tolerability and Efficacy NW-3509A in Patients With Chronic Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Newron Pharmaceuticals SPA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NW-3509A/002/II/2015
Record Dates: First submitted 2015-11-20; First posted 2015-12-08 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Chronic Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NW-3509A (Active Comparator): Patients will start on NW-3509A 15 mg BID and be up-titrated to 20mg, and 25mg BID dependent on tolerability.
  Interventions: Drug: NW-3509A
- Placebo (Placebo Comparator): Patients will receive matching placebo BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NW-3509A — Patients will be given oral doses of 15, 20 and 25 mg BID of NW-3509A
  Arms: NW-3509A
Drug: Placebo — Patients will be given oral dose of matching Placebo
  Arms: Placebo

SUMMARY:
A 4-week Phase IIa study to evaluate the safety and tolerability and efficacy of NW-3509A in patients with chronic schizophrenia that are not responding adequately to their current antipsychotic medication (aripiprazole or risperidone). NW-3509A is given as an oral dose range of 15 to 25 mg, BID in a 1:1 ratio.

DETAILED DESCRIPTION:
This is a prospective, 4-week, randomized, double-blind, placebo-controlled, study designed to evaluate the safety, tolerability, and preliminary efficacy of an oral dose range of NW-3509A of 30 to 50 mg/day (15 to 25 mg, BID) in patients with chronic schizophrenia on a stable dose of an antipsychotic (aripiprazole or risperidone). A minimum of 90 patients will be randomized in a 1:1 ratio to receive either NW-3509A (n=45) or placebo (n=45). Dose increases will be performed only during in-patient setting.

Safety and efficacy assessments will be done on a weekly basis during the randomized treatment period. The assessment of safety will be based on laboratory tests (biochemistry, hematology, and urinalysis), 12-lead standard ECG, vital signs, physical examinations, neurological examinations, C-SSRS, ESRS-A, subjective reporting of any AE by the subject, objective observation of any AE by the Investigator. Pharmacokinetic samples will be taken at various time-points. Efficacy assessments will include the PANSS, CGI-C, CGI-S and the Strauss-Carpenter Level of Functioning (LOF) scale.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female; if female, must not of childbearing potential
2. 18 to 65 years of age, inclusive;
3. Has a current diagnosis of schizophrenia
4. Has a total score on the PANSS < 75.
5. Positive symptoms sub-scale score not to exceed 15; score of ≥4 on no more than 2 positive symptoms
6. Has a Clinical Global Impression - Severity of disease (CGI-S) rating of mildly to moderately severely ill.
7. Is in need of anti-psychotic treatment and is currently receiving a stable dose (minimally for 4 weeks prior to screening of oral risperidone or aripiprazole (at least 2 mg risperidone dose-equivalent).
8. Current symptoms present for at least one month.
9. Patient agrees to be hospitalized for up to 2 days at the start of dosing and at each dose increase

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of NW-3509A in patients with schizophrenia on a stable dose of their current antipsychotic medication (aripiprazole or risperidone). | 27 days
  To evaluate the safety and tolerability of NW-3509A given as an oral dose range of 30 to 50 mg/day (15 to 25 mg, BID) in patients with schizophrenia on a stable dose of their current antipsychotic medication (aripiprazole or risperidone).

SECONDARY OUTCOMES:
Assessment of Positive and Negative Syndrome Scale (PANSS) | 27 days
  Assessment of the PANSS - a 30-item scale designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor attention, and poor impulse control, will be carried out at every visit
Assessment of CGI-S (severity) and CGI-C (change) | 27 days; change from baseline
  Measure of change from baseline will be done at every assessment
Assessment of Strauss-Carpenter Level of Functioning (LOF) scale | 27 days; baseline and end of study
  The LOF scale will be used at baseline and end of study, to evaluate the clinical outcome
Measurement of plasma concentration Cmax | 27 days
  Blood samples will be collected for PK evaluation at time points

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Anand, MD, Study Director — Newron Pharmaceuticals SPA
Locations (5):
- United States (2):
  - Collaborative Neuroscience Network., Garden Grove, California
  - Hassman Research Institute, Berlin, New Jersey
- India (3):
  - KHM Hospital, Chennai, Tamil Nadu
  - Ahana Hospital, Madurai, Tamil Nadu
  - Tirthalli National Institute of Mental Health and Neurosciences, Bangalore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Addington D, Addington J, Maticka-Tyndale E. Assessing depression in schizophrenia: the Calgary Depression Scale. Br J Psychiatry Suppl. 1993 Dec;(22):39-44. PMID 8110442
- [Background] Casey DE, Daniel DG, Wassef AA, Tracy KA, Wozniak P, Sommerville KW. Effect of divalproex combined with olanzapine or risperidone in patients with an acute exacerbation of schizophrenia. Neuropsychopharmacology. 2003 Jan;28(1):182-92. doi: 10.1038/sj.npp.1300023. PMID 12496955
- [Background] Chahine M, Chatelier A, Babich O, Krupp JJ. Voltage-gated sodium channels in neurological disorders. CNS Neurol Disord Drug Targets. 2008 Apr;7(2):144-58. doi: 10.2174/187152708784083830. PMID 18537643
- [Background] Chouinard G, Margolese HC. Manual for the Extrapyramidal Symptom Rating Scale (ESRS). Schizophr Res. 2005 Jul 15;76(2-3):247-65. doi: 10.1016/j.schres.2005.02.013. Epub 2005 Apr 18. PMID 15949657
- [Background] Citrome L. Schizophrenia and valproate. Psychopharmacol Bull. 2003;37 Suppl 2:74-88. PMID 15021863
- [Background] Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0, May 28, 2009 (v4.03 June 14, 2010), U.S. Department of Health and Human Services.
- [Background] Crews KR, Gaedigk A, Dunnenberger HM, Leeder JS, Klein TE, Caudle KE, Haidar CE, Shen DD, Callaghan JT, Sadhasivam S, Prows CA, Kharasch ED, Skaar TC; Clinical Pharmacogenetics Implementation Consortium. Clinical Pharmacogenetics Implementation Consortium guidelines for cytochrome P450 2D6 genotype and codeine therapy: 2014 update. Clin Pharmacol Ther. 2014 Apr;95(4):376-82. doi: 10.1038/clpt.2013.254. Epub 2014 Jan 23. PMID 24458010
- [Background] Goldberg DP, Williams P. A User's Guide to the General Health Questionnaire. 1988. Windsor: NFER-Nelson.
- [Background] Guy W (Ed). Clinical Global Impressions. In ECDEU Assessment Manual for Psychopharmacology, revised, U.S. Department of Health, Education and Welfare Pub. No. (ADM) 76-338. Rockville, MD: NIMH, 1976, 217-222.
- [Background] Kay SR, Fiszbein A, Opler LA. The positive and negative syndrome scale (PANSS) for schizophrenia. Schizophr Bull. 1987;13(2):261-76. doi: 10.1093/schbul/13.2.261. PMID 3616518
- [Background] Lieberman JA, Stroup TS, McEvoy JP, Swartz MS, Rosenheck RA, Perkins DO, Keefe RS, Davis SM, Davis CE, Lebowitz BD, Severe J, Hsiao JK; Clinical Antipsychotic Trials of Intervention Effectiveness (CATIE) Investigators. Effectiveness of antipsychotic drugs in patients with chronic schizophrenia. N Engl J Med. 2005 Sep 22;353(12):1209-23. doi: 10.1056/NEJMoa051688. Epub 2005 Sep 19. PMID 16172203
- [Background] Llerena A, Dorado P, Penas-Lledo EM. Pharmacogenetics of debrisoquine and its use as a marker for CYP2D6 hydroxylation capacity. Pharmacogenomics. 2009 Jan;10(1):17-28. doi: 10.2217/14622416.10.1.17. PMID 19102711
- [Background] Posner K, Oquendo MA, Gould M, Stanley B, Davies M. Columbia Classification Algorithm of Suicide Assessment (C-CASA): classification of suicidal events in the FDA's pediatric suicidal risk analysis of antidepressants. Am J Psychiatry. 2007 Jul;164(7):1035-43. doi: 10.1176/ajp.2007.164.7.1035. PMID 17606655
- [Background] Stingl J, Viviani R. Polymorphism in CYP2D6 and CYP2C19, members of the cytochrome P450 mixed-function oxidase system, in the metabolism of psychotropic drugs. J Intern Med. 2015 Feb;277(2):167-177. doi: 10.1111/joim.12317. PMID 25297512
- [Background] Strauss JS, Carpenter WT Jr. Prediction of outcome in schizophrenia. III. Five-year outcome and its predictors. Arch Gen Psychiatry. 1977 Feb;34(2):159-63. doi: 10.1001/archpsyc.1977.01770140049005. PMID 843175
- [Background] Tiihonen J, Wahlbeck K, Kiviniemi V. The efficacy of lamotrigine in clozapine-resistant schizophrenia: a systematic review and meta-analysis. Schizophr Res. 2009 Apr;109(1-3):10-4. doi: 10.1016/j.schres.2009.01.002. Epub 2009 Jan 30. PMID 19186030
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Zhou SF. Polymorphism of human cytochrome P450 2D6 and its clinical significance: Part I. Clin Pharmacokinet. 2009;48(11):689-723. doi: 10.2165/11318030-000000000-00000. PMID 19817501
- [Background] Zhou SF. Polymorphism of human cytochrome P450 2D6 and its clinical significance: part II. Clin Pharmacokinet. 2009;48(12):761-804. doi: 10.2165/11318070-000000000-00000. PMID 19902987